CLINICAL TRIAL: NCT06976411
Title: Prospective Evaluation for Healing of Iatrogenic Perforation After Repair With Different Materials
Brief Title: Evaluation for Healing of Iatrogenic Perforation After Repair With Different Materials
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mohamed Salah Elwakeel (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Mohamed Salah Elwakeel, Assistant lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-REC 1117 pro
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-12

CONDITIONS: Root Perforation at the Bifurcation Area
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA (Experimental)
  Interventions: Drug: MTA
- Bioceramic (Experimental)
  Interventions: Drug: Bioceramic putty

INTERVENTIONS:
Drug: MTA — Perforation repair using MTA repair material
  Arms: MTA
Drug: Bioceramic putty — Perforation repair using Bioceramic repair material
  Arms: Bioceramic

SUMMARY:
The goal of this clinical trial is to evaluate healing potentiality of MTA and bioceramics materials as a root perforation repair material.

The main questions it aims to answer are:

is there is a significant difference in healing potentiality of MTA and bioceramics materials as a root perforation repair material?

Participants will:

enrollment will be from out-patients clinic of endodontic department, faculty of dentistry, Ain Shams university with root perforations. perforation repair will be done using either bio-ceramic or MTA repair material and preoperative or immediate postoperative CBCT and postoperative CBCT will be taken to compare healing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with root perforation in lower molars.
2. Patients had anon contributory medical history.
3. Patients of age categories between 15 to 50 years old.
4. No sex restriction.
5. Small to medium size perforation.

Exclusion Criteria:

1. Patients with generalized chronic periodontitis.
2. Teeth with difficult isolation.
3. Non restorable teeth.
4. Medically compromised patients.
5. Patients with history of allergies to any of the medications to be used during or after the treatment.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic success in terms of healing | 1 year
  Healing outcome: the presence or absence of lesion and its size were obtained by analyzing CBCT of each case and classified into: Cases with complete resolution of lesion considered as "Healed", reduction of size considered as "Healing", and no size change or increase in lesion size considered as "Failure"
patients with clinical success | 1 year
  A successful clinical outcome was defined as follows: no indication of apical periodontitis, no clinical signs and symptoms, and no loss of function.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry ain shams university, Cairo, Egypt